CLINICAL TRIAL: NCT04206774
Title: BIO|STREAM.ICM France, Submodule of the BIO|STREAM.ICM Registry
Brief Title: BIO|STREAM.ICM France
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS066
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Syncope; Cryptogenic Stroke
MeSH Terms: conditions — Syncope; Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the BIO│STREAM.ICM France submodule is to provide clinical evidence from patients in France on safety and efficacy of the BIOMONITOR system

DETAILED DESCRIPTION:
The BIO|STREAM.ICM submodule will recruit a subset of patients with syncope with uncertain origin and cryptogenic stroke without history of atrial arrhythmia from the existing population enrolled in the BIO|STREAM.ICM registry. The submodule study is designed to provide clinical evidence from patients in France on safety and efficacy of the BIOMONITOR System.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ICM device in accordance with the European guidelines: syncope with uncertain origin or cryptogenic stroke without history of atrial arrhythmia
* Enrolled in the BIO|STREAM.ICM registry

Exclusion Criteria:

* Life-expectancy is less than 3 months
* Already implanted with BIOMONITOR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in French investigation sites, with an indication for Insertable Cardiac Monitors (ICM) in accordance with the European guidelines and followed with the BIOTRONIK Home Monitoring® system.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
SADE free rate | 3 month
  Serious adverse device effect (SADE) free rate related to the BIOMONITOR system

OTHER OUTCOMES:
R-wave amplitude | 3 month
  Assessment of R-wave Amplitude (Millivolt) detected by the BIOMONITOR and transmitted via Home Monitoring
Noise burden | 3 month
  Assessment of electrical noise burden (%) detected by the BIOMONITOR and transmitted via Home Monitoring
Ventricular rate | 3 month
  Assessment of mean ventricular rate (bpm) detected by the BIOMONITOR and transmitted via Home Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Romain ESCHALIER, Pr., Principal Investigator — Hôpital Gabriel Montpied
Locations (3):
- France (3):
  - Hôpital Gabriel Montpied, Clermont-Ferrand, Caen
  - CH Villefranche Sur Saone, Gleizé
  - CHRU de Tours, Hopital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: No